CLINICAL TRIAL: NCT06520839
Title: Genetic Factors of Erectile Dysfunction Degree and Response to Tadalafil Treatment in Patients With Diabetes
Acronym: EDGEN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Boštjan Hostnik, MD, internal medicine physician, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Erectile Dysfunction With Diabetes Mellitus
Keywords: Erectile Dysfunction; Diabetes Mellitus
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with diabetes and erectile dysfunction (Experimental): We will include in the study 90 patients with diabetes and erectile dysfunction. We will use the IIEF-5 questionnaire to confirm the diagnosis of erectile dysfunction. Patients between the ages of 40 and 65 who score 21 points or less on the IIEF-5 scale will be included in the study. Each patient will receive drug tadalafil 5 mg every day for three months.
  Interventions: Drug: Tadalafil 5mg

INTERVENTIONS:
Drug: Tadalafil 5mg — We will include in the study 90 patients with diabetes and erectile dysfunction. We will use the IIEF-5 questionnaire to confirm the diagnosis of erectile dysfunction. Patients between the ages of 40 and 65 who score 21 points or less on the IIEF-5 scale will be included in the study. Each patient will receive drug tadalafil 5 mg every day for three months.
  Other Names: Tadilecto 5 mg

SUMMARY:
The goal of this clinical trial is to examine the genetic markers of erectile dysfunction degree in patients with diabetes and find new predictive models based on genetic factors, with which we will be able to more accurately address the adequacy of treatment in patients with diabetes, and thus have a long-term impact to reduce side effects of treatment. We will look for a predictive model based on genetic analysis to determine in the future patients with a good response to treatment with phosphodiesterase type 5 inhibitors, in our case tadalafil 5 mg daily. The main questions it aims to answer are:

1. Genetic alterations in the NO signaling pathway affect the degree of erectile dysfunction and the response to tadalafil treatment in patients with diabetes.
2. Genetic alterations in the folate pathway affect the degree of erectile dysfunction and the response to tadalafil treatment in patients with diabetes.
3. Genetic factors of the vascular wall influence the degree of erectile dysfunction and the response to tadalafil treatment in patients with diabetes.
4. Genetic changes in the pathways of tadalafil metabolism and action influence the response to the treatment of erectile dysfunction in patients with diabetes.

Participants will take the drug tadalafil 5 mg every day for three months. The level of erectile dysfunction will be assessed with the IIEF-5 questionnaire at the beginning of the study and after three months of taking the drug.

DETAILED DESCRIPTION:
We will include in the study 90 patients with diabetes and erectile dysfunction. We will use the IIEF-5 questionnaire to confirm the diagnosis of erectile dysfunction. Patients between the ages of 40 and 65 who score 21 points or less on the IIEF-5 scale will be included in the study.

The research will be clinically pharmacological, prospective, interventional and genetic-associative. Patients will be selected sequentially, according to their willingness to participate in the research, taking into account the inclusion and exclusion criteria. As a result, they will not be subject to randomization. At the first examination and after signing the informed consent form for participation in the research, blood will be taken from the patients for laboratory and molecular genetic tests, they will receive the drug for the treatment of erectile dysfunction tadalafil, which they will receive in a dose of 5 mg daily for a period of three months . After three months, patients will complete the IIEF-5 questionnaire again.

At the beginning of the research, we will explain the course and purpose of the research to the people involved, they will fill out a consent form for participating in the research. Upon inclusion, we will perform the following on all subjects:

* History and clinical examination (including weight, height and body mass index). The degree of erectile dysfunction will be classified using the IIEF-5 questionnaire into four categories, namely severe (5-7 points), moderate (8-11 points), mild to moderate (12-16 points) and mild form (17-21 points ) of erectile dysfunction.
* Laboratory tests Peripheral venous blood will be taken to determine laboratory parameters: renal function, hepatogram, lipidogram, HbA1c (TIR), PSA, TSH, LH, FSH, PRL, SHBG, testosterone (total and free), folic acid.
* Molecular genetic tests 3-5 ml of peripheral venous blood will be taken from the examinees in a test tube with EDTA. Centrifugation will separate the blood plasma from the cellular part of the blood. Genomic DNA will be isolated from the cellular part of the blood using commercial reagent sets (DNA Mini Kit and Flexigene DNA kit; Qiagen, Hilden, Germany). To determine polymorphisms of individual nucleotides in the genes of the synthesis pathway, NO function and folate pathway, we will use modern high-throughput methods based on the real-time PCR reaction, such as the 5'-exonuclease test (TaqMan SNP genotyping assay; Applied Biosystems, Foster City, CA , USA) and allele-specific competitive PCR reactions (KASPar assay; KBiosciences, Herts, UK).

Candidate genes were selected based on a literature review, focusing on pathways related to the molecular pathogenesis of erectile dysfunction and pathways related to the metabolism and action of tadalafil. Based on a review of the databases (dbSNP, PharmGKB) and the literature, we searched for genetic changes in the mentioned genes that are common in the white race and affect the expression of the gene or the function of the written protein. Based on this, we decided to include the following genes and polymorphisms in the analysis:

* signaling pathway NO: NOS3: 894G/T (rs1799983), 786T/C (rs2070744)
* vascular wall factors: VEGF: 460T/C (rs833061), 1154G/A (rs1570360), 2578A/C (rs699947); ACE: rs1800764, rs4343, rs1799752; ACE2: rs2285666, rs1978124
* folate pathway: MTHFR: rs1801133 (p.Ala222Val; c. 677 C>T), rs1801131 (p.Glu429Ala; c.1298 A>C), MS: rs1805087 (p.Asp919Gly; c.2756A>G), MTRR : rs1801394 (p.Ala66Gly; 66A>G)
* tadalafil metabolism: CYP3A4*22 and CYP3A5*3
* tadalafil target: PDE5A: rs12646525, rs3806808

ELIGIBILITY:
Inclusion Criteria:

* We will include in the study 90 patients with diabetes and erectile dysfunction. We will use the IIEF-5 questionnaire to confirm the diagnosis of erectile dysfunction. Patients between the ages of 40 and 65 who score 21 points or less on the IIEF-5 scale will be included in the study.

Exclusion Criteria:

* patients receiving any form of organic nitrate in regular therapy or as necessary due to ischemic heart disease, patients who have already suffered a cardiovascular event (heart attack, stroke, manifest peripheral arterial disease), users of illegal drugs, alcoholics, demented patients , patients with psychiatric diseases, patients with pancreatogenic form of diabetes, patients with glucocorticoids and immunosuppressants induced form of diabetes and patients with monogenic form of diabetes. Patients with hypogonadism, prostate malignancy, patients with a psychogenic form of erectile dysfunction, patients with premalignant and malignant genital lesions, patients with Peyronie's disease, patients after injury, surgery and radiation in the pelvic area and patients with congenital diseases of the penis will also be excluded from the research. We will also exclude from the research patients who withdraw from participation in the research during the research for personal or any other reasons.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Genetic alterations in the NO signaling pathway affect the degree of erectile dysfunction and the response to tadalafil treatment in patients with diabetes. | 3 months
  Genetic polymorphisms
Genetic variations in the folate pathway influence the degree of erectile dysfunction and the response to tadalafil treatment in patients with diabetes. | 3 months
  Genetic polymorphisms
Vascular wall genetic factors influence the degree of erectile dysfunction and the response to tadalafil treatment in patients with diabetes. | 3 months
  Genetic polymorphisms
Genetic variations in tadalafil metabolism and action pathways influence response to erectile dysfunction treatment in patients with diabetes. | 3 months
  Genetic polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: Boštjan Hostnik, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No